**IRAS ID:** 

**Trial Name:** 



320293



## **Participant Informed Consent Form**

**Evaluation of Pilot Online Binge Eating Disorder Group in under 18s.** 

| Chief<br>Investigator:<br>Principal<br>Investigator:<br>Participant Ide<br>number: | | Dominique Muhumuza Dominique Muhumuza entification | | |
|---|---|---|---|---|
| 1. | I confirm that I have: | | | |
| • | <ul> <li>read and understand the information sheet PIS Service User - BE Group Intervention<br/>2022.docx for the above study.</li> </ul> | | | |
| • | <ul> <li>had enough time to think whether or not I want to take part, ask questions and get answers that I think are reasonable.</li> </ul> | | | |
| • | <ul> <li>understood that this study is designed to further scientific knowledge and that all procedures<br/>have been approved by the Research Ethics Committee of Newman University and Research<br/>Ethics Committee of Coventry Warwickshire Partnership NHS Trust.</li> </ul> | | | |
| 2. | <ol> <li>I understand that my taking part is voluntary and that I am free to stop taking part at any time<br/>without giving any reason, without my medical care or legal rights being affected.</li> </ol> | | | |
| 3. | 3. I agree to try and complete the questionnaires. I understand that I can take a break or stop completing them if I wish. | | | |
| 4. I understand that: | | | | |
| • | I am partici | pating in a group | | |
| • | • I will be asked to complete weekly tasks as part of the group intervention | | | |
| • | My parent vintervention | will be asked to attend an informati<br>า | on session to s | upport me through this group |
| 5. | . I understand that my questionnaires and feedback may be looked at by people from the Coventry and Warwickshire Partnership trust or Newman University. I give permission for these individuals to have access to all information collected. | | | |
| 6. | . I agree that my carer, friend or relative may be asked questions about my treatment | | | |
| 7. | I understand that information collected will be kept confidential. However, if I tell the researchers something they think is likely to result in immediate harm to myself or others, they may have to talk to me about disclosing this in line with the law and local safeguarding procedures. | | | |
| 8. | I agree the | ED team to inform my GP that I ar | m participating i | in this project. |
| 9. | I agree to t | take part in the above study. | | |
| You | r name (in d | capitals) | Date | Signature |
| Nam | e of persor | n taking consent (in capitals) | Date | Signature |
| | | n recording consent (if different) | Date | Signature |
| (III C | apitals) | | | |

When completed, the original should be kept in the Investigator Site File, a copy should be given to the patient and one kept in the study notes along with the Participant Information Sheet.